CLINICAL TRIAL: NCT06646861
Title: Head and Neck Cancer Rehabilitation: the CaRe Feasibility Study
Acronym: CaRe
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Irish Cancer Society (Other); St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Grainne Sheill, Adjunct Assistant Professor, University of Dublin, Trinity College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2247
Record Dates: First submitted 2024-10-11; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-09

CONDITIONS: Head and Neck Cancer Survivors
Keywords: Exercise; Rehabilitation; Survivorship
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise (Experimental): Multi-modal exercise programme The 10-week multi-modal exercise programme will comprise of twice weekly online supervised group-based exercise sessions. Each exercise session will last approximately 1 hour and consist of a combination of aerobic, resistance and balance and flexibility exercises.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — A combination of aerobic, resistance, balance and flexibility exercises will be included.

SUMMARY:
Introduction: As both the number of cancer survivors and the length of survival time are increasing, long-term health issues related to cancer and its treatment are becoming more prevalent. Research suggests that exercise can mitigate a number of negative health consequences of head and neck cancer and improve physical function and quality of life. Multi-modal exercise interventions have been proposed as a cornerstone for survivorship care. However, studies evaluating exercise programmes in head and neck cancer populations are lacking.

Purpose: To evaluate the feasibility and acceptability of a multi-modal exercise rehabilitation programme for survivors of head and neck cancer in a real-world, standard practice setting.

Methods and analysis: In this single-arm prospective feasibility study, survivors of head and neck cancer (n=29) will undergo a 10-week multi-modal exercise programme. The study population will comprise of cancer survivors attending outpatient services in an Irish national cancer centre. Participants will be aged 18 or older and have completed treatment with curative intent.

Feasibility will be evaluated in terms of recruitment, adherence and compliance to the programme. Secondary outcomes will examine physical function and quality of life measures. In addition, the acceptability of the programme will be assessed through patient feedback.

Ethics and dissemination: Ethical approval is pending from the St. James's Hospital and Tallaght University Hospital Research and Ethics Committee. The study results will be used to optimise the intervention content, and may serve as the foundation for a larger definitive trial. Results will be disseminated through peer-review journals, congresses and relevant clinical groups.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Over 18 years old
* In the first two years after treatment for head and neck cancer
* Medically fit to participate in low to moderate physical activity

Exclusion Criteria:

* Individuals with moderate or severe cognitive impairment
* Pregnancy
* Receiving treatment in the palliative setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Programme feasibility | From enrolment until end of study intervention at 10 weeks
  Recruitment rates (percentage of eligible study population that consented to participation), programme adherence (number of prescribed supervised and unsupervised sessions completed), retention, acceptability of the intervention and adverse events. Reasons for attrition or non-compliance will be identified through qualitative evaluation with participants.

SECONDARY OUTCOMES:
The Neck Disability Index | From enrolment until end of study intervention at 10 weeks
  The Neck Disability Index will assess neck pain.
Quality of Life | From enrolment until end of study intervention at 10 weeks
  The functional assessment of cancer therapy head and neck questionnaire will be used to measure quality of life.
  The higher the score, the better the QOL.
Physical Function | From enrolment until end of study intervention at 10 weeks
  The 30 second Sit to Stand test, hand grip strength and clinical frailty scale. 30 second Sit to Stand: higher score associated with better outcomes Hand Grip Strength: higher score associated with better outcomes Clinical Frailty Scale: Lower values are associated with better outcomes
Physical Activity | From enrolment until end of study intervention at 10 weeks
  Self-reported physical activity will be collected using the Godin Leisure-Time Physical Activity Questionnaire.
  The GLTEQ is a 4-item self-administered questionnaire with the first three questions seeking information on the number of times one engages in mild, moderate and strenuous activity in bouts of at least 15 min duration in a typical week. Total leisure activity score is then calculated based on number of bouts at each intensity multiplied by 3, 5, and 9 metabolic equivalents and summed. A higher score means more physically active.
Cancer Related Fatigue | From enrolment until end of study intervention at 10 weeks
  Brief Fatigue Inventory This 9-item scale assesses the severity and interference of fatigue based on a 0 (no fatigue) to 10 (greatest fatigue) scale
Oral Intake | From enrolment until end of study intervention at 10 weeks
  The Functional Oral Intake Scale This scale reflects the functional oral intake of patients (1-7) where 7 indicates no restrictions to oral intake and better outcomes
Lymphoedema | From enrolment until end of study intervention at 10 weeks
  Lymph Scanner

CONTACTS AND LOCATIONS:
Overall Officials: Grainne Sheill, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- School of Medicine, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided